CLINICAL TRIAL: NCT04278092
Title: Paclitaxel Plus Cetuximab for the Treatment of Recurrent and/or Metastatic Head and Neck Cancer After First-line Checkpoint Inhibitor Failure: A Multicenter, Single Arm Study
Brief Title: Paclitaxel Plus Cetuximab After First-line Checkpoint Inhibitor Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Thorsten Fuereder, Assoc.Prof., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PACE ACE
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Paclitaxel; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Paclitaxel plus Cetuximab (Experimental): Paclitaxel combination with weekly cetuximab will be administered for up to six cycles. Thereafter weekly cetuximab maintenance will be given.
  Interventions: Drug: Paclitaxel; Drug: Cetuximab

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel 175 mg/m2, q21
  Other Names: Taxol
Drug: Cetuximab — Cetuximab 400mg/m2 loading dose followed by weekly 250mg/m2
  Other Names: Erbitux

SUMMARY:
Immune checkpoint inhibitors (CPI) such as pembrolizumab or nivolumab have been recently approved for the treatment of recurrent/metastatic head and neck cancer (HNSCC). However, only a minority of patients respond to therapy. From the clinical point of view the optimal management of patients progressing on or after CPI therapy is still a challenge. Retrospective analysis showed that HNSCC patients, who progressed on/after CPI, demonstrated an overall response rate (ORR) of up to 30% subsequent to chemotherapy +/- cetuximab treatment. It is the aim of this study to evaluate if paclitaxel plus cetuximab after first line pembrolizumab failure is an effective salvage therapy in 50 R/M HNSCC patients. The primary endpoint is ORR according to RECIST V 1.1.

ELIGIBILITY:
Inclusion Criteria:

* The patient has provided written informed consent prior to any study-related procedure.
* The patient is at least 18 years of age
* Histologically proven locally advanced unresectable, recurrent and/or metastatic squamous cell carcinoma of the oropharynx, hypopharynx, larynx or oral cavity not amenable for salvage surgery
* p16 status has to be determined for oropharyngeal carcinomas
* Documented progressive disease based on investigator assessment according to RECIST 1.1, following receipt of a pembrolizumab based regimen given as first line therapy for R/M SCCHN
* Measurable disease according to RECIST 1.1.
* The patient has a life expectancy of at least 3 months.
* Has a performance status of ≤ 2 on the ECOG Performance Scale
* Female patient of childbearing potential should have a negative urine or serum pregnancy prior to study . If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female patients of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study until 120 days after the last dose of study medication. Patients of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male patients should agree to use an adequate method of contraception starting with the first dose of study therapy until 120 days after the last dose of study therapy.
* Demonstrate adequate organ function as defined in table 1, all screening labs should be performed within 14 days of treatment initiation.

Exclusion Criteria:

* Prior taxane therapy is not allowed except as part of induction therapy for locally advanced disease (completed at least 6 months before study entry)
* Prior cetuximab therapy is not allowed except as part of either induction therapy or in combination with radiotherapy treatment for locally advanced disease (completed at least 6 months before study entry)
* Patients with nasopharyngeal carcinomas or salivary glands cancers
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency including a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis A/B or Hepatitis C
* Has had prior pembrolizumab within 2 weeks prior to study day 1 or who has not recovered (i.e., recovery to ≤ Grade 1 or baseline grade prior to pembrolizumab) from (immune- related) adverse events other than endocrine side effects.
* Has had prior chemotherapy or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., recovery to ≤ Grade 1 or baseline grade prior to pembrolizumab) from adverse events due to a previously administered agent.
* Has had chemotherapy, targeted therapy or investigational drugs after checkpoint inhibitor failure for second line therapy .
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit until 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 3 months
  To evaluate the Overall Response Rate (CR/PR) rate according to RECIST V 1.1

SECONDARY OUTCOMES:
Median Overall Survival | 2 years
  The interval between start of treatment and death from any cause
Median Progression Free Survival | 2 years
  The interval between start of treatment and date of progression, or death, from any cause
Median Duration of response | 2 years
Health-related quality-of-life scores per patient measured according to the European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) C-30 scoring manual | 2 years
Health-related quality-of-life scores per patient measured according to the European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) H&N35 scoring manual | 2 years
Number of participants with adverse events | 2 years
  AEs, treatment-related AEs, serious adverse events (SAEs), and treatment-related SAEs will be tabulated using worst grade per NCI CTCAE v 5.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Fuereder, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria